CLINICAL TRIAL: NCT04849195
Title: Comparison of Different Feature Engineering Methods for Automated ICD Coding
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: Sponsor
Other Study IDs: 2021-1425-02
Record Dates: First submitted 2021-04-13; First posted 2021-04-19 (Actual); Last update posted 2021-04-19 (Actual); Status verified 2021-04

CONDITIONS: Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Model training and test group: Data set will be split into training group and test group, where training group will be used for model building, and test group for subsequent evaluation and verification.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Using traditional machine learning classifiers, this study targets on comparing bag-of-words, word2cec and roberta on automated ICD coding related to cardiovascular diseases in Chinese corpus.

DETAILED DESCRIPTION:
ICD coding is quite important as it serves as basis for a wide range of economic and academic applications. Currently, manual coding is mainly adopted, which faces several limits like being time-consuming and prone to error, and this makes automated ICD coding via machine learning a hot research topic.

As an inevitable phase during machine learning, feature engineering plays a crucially important role in leading to promising coding performance. Although have reached enlightening conclusions, existing studies lacked comparison of different feature engineering methods. Finding out what methods under what circumstances perform better can be quite helpful in promoting practical applications of automated coding.

The investigators will implement this study based on inpatient' data collected from electronic medical records from Fuwai Hospital, the world's largest medical center for cardiovascular disease. Bag-of-words, word2cec and roberta will be respectively used to extracted features from training data. Then code-wise logistic regression classifiers and support vector machine classifiers will be trained to auto-assign codes. Afterwards, performances of the models on test data will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Admissions in Fuwai Hospital, from January 1, 2019, to February 28, 2019

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Admissions in Fuwai Hospital
Sampling Method: Non-Probability Sample
Enrollment: 6947 (Estimated)
Dates: Start 2021-03-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
ICD-10 codes for each admission | At the end of enrollment
  Each admission will be a sample in this study. The ICD-10 codes assigned by medical coders for each admission will be collected as the primary outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Wei Zhao, PhD, Principal Investigator — China National Center for Cardiovascular Diseases
Locations (1):
- Fuwai Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No